CLINICAL TRIAL: NCT03963206
Title: CLERANCE HCC, Cabozantinib toLERANCE Study in HepatoCellular Carcinoma
Brief Title: Cabozantinib toLERANCE Study in HepatoCellular Carcinoma (CLERANCE)
Acronym: CLERANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0977; 2019-001142-18 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Cabozantinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib group (Other): patients will receive Cabozantinib (within the framework of its MA) (an ECG is added)
  Interventions: Drug: Cabozantinib group

INTERVENTIONS:
Drug: Cabozantinib group — The patient starts at 60 mg / day at a distance from meals In the event of intolerance to this dose of 60 mg; specific adapted measures will be taken according to the recommendations of the good practices of use of Cabozantinib within the framework of its MA. If the symptomatic treatments are not enough, each investigator can adapt the dose of Cabozantinib reducing it to 40 or even 20 mg / day Cabozantinib will be continued for as long as radiological and / or clinical benefit is observed for the patient (no progression of the disease) or until the occurrence of unacceptable toxicity.

SUMMARY:
Hepatocellular carcinoma (HCC) is a common tumor (the 8th leading cause of cancer in France) and has a poor prognosis. It is the 3rd leading cause of cancer deaths in the world. In the early stages (low tumor mass), HCC can be treated for curative purposes by surgical resection, percutaneous ablation or liver transplantation. When the tumor mass is larger (> 3 nodules) but remains confined to the liver, the standard treatment is hepatic intra-arterial chemoembolization (TACE). In the event of failure of the latter or if the tumor dissemination progresses in the portal venous system or in the form of metastases, the systemic treatments are then indicated.

In 1st line, the reference treatment is a tyrosine kinase inhibitor (ITK) Sorafenib.

Cabozantinib obtained the European and French authorization (AMM) in November 2018 for its use in case of failure of Sorafenib in patients with HCC.

The main objective is the evaluation of the safety of Cabozantinib administered to patients with intermediate HCC ineligible for chemoembolization or advanced HCC after failure of Sorafenib and possibly another systemic anticancer line.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age ≥ 18 years).
* Patient with a histologically proven HCC, or by radiology if cirrhotic liver (according to international recommendations).

Patient with stage B BCLC classification after failure or impossibility of transarterial chemoembolization (TACE), or advanced stage C having already received one to two systemic lines, including one by Sorafenib.

* eastern cooperative oncology group score of 0 or 1 (ECOG).
* Child-Pugh A5 or A6 score.
* Disease evaluable by RECIST v1.1 and mRECIST.
* Hemoglobin> 8.5g / dL.
* Platelets> 60 giga / L.
* neutrophils> 1.2 giga / L.
* ALAT and ASAT <5N
* Patient having a normal magnesium level
* Clearance with creatinine> 40ml / min (by the MDRD formula).
* For patients who have had radiotherapy on the liver: a wash out of at least one month before the start of the treatment under study must be respected.
* For patients who have had a radioembolization a wash out of at least three months before the beginning of the treatment under study must be respected.
* Patient who agreed to participate in the study and signed the informed consent.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient with another cancer not cured or whose complete remission has been obtained for less than 2 years compared to the date of inclusion in CLERANCE.
* Patients eligible for surgical resection or radiofrequency ablation or liver transplantation or TACE according to international recommendations.
* Patient who has already had more than two lines of systemic treatment for his HCC (tyrosine kinase inhibitor, intravenous cytotoxic chemotherapy, immunotherapy, hormonal therapy for HCC).
* Patient who has never received Sorafenib in his previous systemic line (s).
* Patient who has already received a c-MET inhibitor.
* Patient with chronic viral B infection known not treated with a nucleoside / nucleotide analogue.
* Patients infected with HIV known (even if it is viro-suppressed by anti-retroviral treatments).
* Patients with or at risk for severe bleeding (a gastroscopy should be performed every two years if the patient doesn't have varicose veins and every year if the patient has varicose vein).
* Patients with inflammatory bowel diseases (Crohn's disease, ulcerative colitis, peritonitis, diverticulitis, appendicitis)
* Patient with galactose intolerance or Lapp lactase deficiency, or glucose or galactose malabsorption syndrome.
* Patients with tumor infiltration of the digestive tract with risk of fistulation
* Patients with recent digestive surgery (<1 month) or not yet fully healed.
* Patients with QTcF> 480 ms on inclusion ECG.
* Known hypersensitivity to Cabozantinib or to any of the excipients.
* Pregnant or nursing woman.
* Patient of childbearing age without mechanical contraception.
* Patient placed under safeguard of justice (tutelage or curatorship).
* Patient not benefiting from social security.
* Patient participating in another interventional research in progress or including an exclusion period still in progress at pre-inclusion (except interventional research with minimal risks and constraints that do not interfere with the judgment criteria of the study according to the judgment of the coordinating investigator).

Chronic active C infection is not a contraindication. Treatment with direct antiviral agents is left to the discretion of each investigator, but the viremic or cured status of each patient should be mentioned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
survival of the patient after start of treatment | Year 1
  Overall Survival (OS) defined as the time (in months) between the start of treatment with Cabozantinib and the date of death from all causes; patients who are alive or lost to follow-up at the time of the analysis will be censored on the last follow-up date

SECONDARY OUTCOMES:
dosage modification for adverse effect | Year 1
  Incidence of changes in the dose of Cabozantinib for adverse effect during treatment (including daily dose reductions, dose spacings, discontinuation and permanent cessation of treatment for intolerance).
Daily median dose of Cabozantinib | Year 1
  Daily median dose of Cabozantinib calculated between the start of treatment with Cabozantinib and the day of final cessation (including death)
Number of patients with each dose of Cabozantinib | Year1
  calculation of the number of patients with a dose of Cabozantinib 60 mg, 40 mg or 20 mg at the end of treatment or at the end of the study.

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens Picardie - Hôpital Sud, Amiens
  - CHU Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier de Boulogne sur mer, Boulogne-sur-Mer
  - Centre hospitalier universitaire Côte de nacre, Caen
  - Hôpital Beaujon, Clichy
  - CHRU de Lille-Hôpital Claude Huriez, Lille
  - CHU Dupuytren, Limoges
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon
  - APHM - Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - APHP - Hôpital St Antoine, Paris
  - Hôpital haut- lévêque, Pessac
  - Hôpital Robert Debré - CHU de Reims, Reims
  - CHRU Rennes site pontchaillou, Rennes
  - CHU de St Etienne, Saint-Priest-en-Jarez
  - CHU Toulouse PURPAN, Toulouse
  - Hôpital Brabois adulte - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] P Merle - Cabozantinib toLERANCE Study in HepatoCellular Carcinoma - Liver Cancer (Publication in progress)